CLINICAL TRIAL: NCT02143934
Title: Host and Parasites Factors Contributing to Risk of Plasmodium Re-infection and Morbidity in Elementary School Children in Maprik, East Sepik Province
Brief Title: Effect of Liver and Blood-stage Treatment on Subsequent Plasmodium Reinfection and Morbidity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Papua New Guinea Institute of Medical Research (Other Government)
Collaborators: Walter and Eliza Hall Institute of Medical Research (Other); Swiss Tropical & Public Health Institute (Other); Barcelona Centre for International Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 07200734
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Plasmodium Vivax Infection; Plasmodium Vivax Clinical Episode; Plasmodium Falciparum Infection; Plasmodium Falciparum Clinical Episode
Keywords: Plasmodium vivax; Hypnozoites; Primaquine; Liver-stage; Blood-stage; Plasmodium falciparum
MeSH Terms: conditions — Malaria, Vivax; Malaria, Falciparum | interventions — Primaquine; Chloroquine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primaquine (Active Comparator): Primaquine, 0.5mg/kg/day, 20 days directly observed treatment Chloroquine, 25mg/kg total dose, divided over 3 days directly observed treatment Artemether-Lumefantrine, 3 days BD
  Interventions: Drug: Primaquine; Drug: Chloroquine; Drug: Artemether Lumefantrine
- Placebo (Placebo Comparator): Placebo, 20 days directly observed treatment Chloroquine, mg/kg, 3 days directly observed treatment Artemether-Lumefantrine, 3 days BD
  Interventions: Drug: Placebo; Drug: Chloroquine; Drug: Artemether Lumefantrine

INTERVENTIONS:
Drug: Primaquine
  Arms: Primaquine
Drug: Placebo — Sugar pills, appearance identical to Primaquine tablets
  Arms: Placebo
Drug: Chloroquine
Drug: Artemether Lumefantrine
  Other Names: Coartem

SUMMARY:
This study specifically seeks to quantify the contribution of relapes to the burden of P. vivax infections and disease by determining on the effect of radical pre-erythrocytic and erythrocytic clearance on subsequent rates of Plasmodium spp. infection and disease in children aged 5-10 years in a treatment to re-infection study design. In order the clear liver-stage/blood-stages G6PD-normal children were randomised to receive Chloroquine (3 days, standard dose) and Coartem (3 days, standard dose) plus either i) primaquine (20 days, 0.5mg/kg) or ii) placebo (20days). These drugs were administered over a period of 4 weeks.

In addition to this epidemiological data, the study will assess the natural acquisition of cellular and humoral immune responses to P. falciparum and P. vivax, thus assisting in the determination of correlates of clinical immunity to P. falciparum and P. vivax in PNG children aged 5-10 years.

These data will not only be essential for development of future vaccines against P. vivax and P falciparum but provide invaluable insight into the contribution of long-lasting liver-stages to the force of infection with P. vivax that will contribute towards designing more rational approaches to the treatment of P. vivax both in the context of case management and future attempts at elimination.

ELIGIBILITY:
Inclusion Criteria:

* aged 5-10 years (±3 months)
* permanent residents of the area
* absence of history of hypersensitivity reactions to the drugs

Exclusion Criteria:

* chronic illness
* severe malnutrition (weight-for-age nutritional Z score [WAZ] <60th percentile)
* severe anemia (Hb <5 g/dL),
* G-6-PD deficiency (<60% G-6-PD activity)
* permanent disability, which prevents or impedes study participation. Any 1 or more of the criteria is sufficient to exclude study participation.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 524 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Time to first or only Plasmodium vivax infection by light microscopy and PCR | 8 months post-baseline
Time to first or only clinical P. vivax episode | 8 months post-baseline

SECONDARY OUTCOMES:
Time to first or only P. falciparum infection by light microscopy and PCR | 8 months post-baseline
Time to first or only P. ovale infection by light microscopy and PCR | 8 months post-baseline
Time to first or only P. malariae infection by light microscopy and PCR | 8 months post-baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ivo Mueller, PhD, Principal Investigator — Walter and Eliza Hall Institute of Medical Research; Centre de Recerca en Salut Internacional de Barcelona (CRESIB); Inoni Betuela, MD PhD, Principal Investigator — PNG Institute of Medical Research; Louis Schofield, PhD, Principal Investigator — Walter and Eliza Hall Institute of Medical Research
Locations (1):
- PNG Institute of Medical Research, Maprik, East Sepik Province, Papua New Guinea

REFERENCES:
- [Derived] Potter GE, Callier V, Shrestha B, Joshi S, Dwivedi A, Silva JC, Laurens MB, Follmann DA, Deye GA. Can incorporating genotyping data into efficacy estimators improve efficiency of early phase malaria vaccine trials? Malar J. 2023 Dec 19;22(1):383. doi: 10.1186/s12936-023-04802-0. PMID 38115002
- [Derived] Potter GE, Callier V, Shrestha B, Joshi S, Dwivedi A, Silva JC, Laurens MB, Follmann DA, Deye GA. Can incorporating genotyping data into efficacy estimators improve efficiency of early phase malaria vaccine trials? Res Sq [Preprint]. 2023 Sep 22:rs.3.rs-3370731. doi: 10.21203/rs.3.rs-3370731/v1. PMID 37790581
- [Derived] Stadler E, Cromer D, Mehra S, Adekunle AI, Flegg JA, Anstey NM, Watson JA, Chu CS, Mueller I, Robinson LJ, Schlub TE, Davenport MP, Khoury DS. Population heterogeneity in Plasmodium vivax relapse risk. PLoS Negl Trop Dis. 2022 Dec 19;16(12):e0010990. doi: 10.1371/journal.pntd.0010990. eCollection 2022 Dec. PMID 36534705
- [Derived] Holzschuh A, Gruenberg M, Hofmann NE, Wampfler R, Kiniboro B, Robinson LJ, Mueller I, Felger I, White MT. Co-infection of the four major Plasmodium species: Effects on densities and gametocyte carriage. PLoS Negl Trop Dis. 2022 Sep 13;16(9):e0010760. doi: 10.1371/journal.pntd.0010760. eCollection 2022 Sep. PMID 36099312
- [Derived] Hofmann NE, Karl S, Wampfler R, Kiniboro B, Teliki A, Iga J, Waltmann A, Betuela I, Felger I, Robinson LJ, Mueller I. The complex relationship of exposure to new Plasmodium infections and incidence of clinical malaria in Papua New Guinea. Elife. 2017 Sep 1;6:e23708. doi: 10.7554/eLife.23708. PMID 28862132
- [Derived] Wampfler R, Hofmann NE, Karl S, Betuela I, Kinboro B, Lorry L, Silkey M, Robinson LJ, Mueller I, Felger I. Effects of liver-stage clearance by Primaquine on gametocyte carriage of Plasmodium vivax and P. falciparum. PLoS Negl Trop Dis. 2017 Jul 21;11(7):e0005753. doi: 10.1371/journal.pntd.0005753. eCollection 2017 Jul. PMID 28732068
- [Derived] Robinson LJ, Wampfler R, Betuela I, Karl S, White MT, Li Wai Suen CS, Hofmann NE, Kinboro B, Waltmann A, Brewster J, Lorry L, Tarongka N, Samol L, Silkey M, Bassat Q, Siba PM, Schofield L, Felger I, Mueller I. Strategies for understanding and reducing the Plasmodium vivax and Plasmodium ovale hypnozoite reservoir in Papua New Guinean children: a randomised placebo-controlled trial and mathematical model. PLoS Med. 2015 Oct 27;12(10):e1001891. doi: 10.1371/journal.pmed.1001891. eCollection 2015 Oct. PMID 26505753